CLINICAL TRIAL: NCT03428542
Title: The Effects of Yoga on Psychological and Physiological Health in a Population Based Cohort
Brief Title: Yoga and Psychological and Physiological Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Olle Melander, Professor, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015610
Record Dates: First submitted 2018-01-30; First posted 2018-02-09 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Stress; Anxiety; Depression; Sleep; Physiological Stress
Keywords: yoga; stress; anxiety; depression; sleep quality; physiological stress; biomarkers
MeSH Terms: conditions — Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Parallel-group RCT with three arms during 5 weeks. Subjects were randomized to a control group, the Yin Yoga intervention group or the YOMI intervention group. YOMI intervention combines Yin yoga with psychoeducation and mindfulness practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (No Intervention): Instructed not to practice any yoga or mindfulness during the five-week study period.
- Yin yoga intervention arm (Active Comparator): The Yin yoga intervention arm will receive Yin yoga, a calm-paced practice that uses seated and lying down positions.
  Participants were also provided a CD which contained a 10-minute voice recording called conscious breathing. The guided instructions encouraged participants to keep awareness on their breath and to use calm, slow, nostril breathing.
  Interventions: Behavioral: Yin yoga
- YOMI program intervention arm (Active Comparator): The YOMI intervention arm will receive stress education + yoga, and bring together education about stress, mindfulness and yoga practice. It will involve weekly group meetings, homework, and yoga postures. Stress education and mindfulness will make up one portion of the intervention. This will take place in a group lecture format and shall be conducted by a mental health professional(s). Yoga practice in a group format will make up the second portion of the intervention.
  Participants were also provided a CD which contained a 10-minute voice recording called conscious breathing. The guided instructions encouraged participants to keep awareness on their breath and to use calm, slow, nostril breathing.
  Interventions: Behavioral: YOMI

INTERVENTIONS:
Behavioral: Yin yoga — Yin yoga 2 times per week for 5 weeks. Daily breathing assignments.
  Arms: Yin yoga intervention arm
Behavioral: YOMI — 30 minutes of psychoeducation combined with mindfulness practice followed by 60 minutes of Yin yoga allowing the psychological theme to be further explored, aided by verbal instructions of the yoga teacher. 2 times per week for 5 weeks.
  Daily breathing assignments.
  Arms: YOMI program intervention arm

SUMMARY:
This study aims to evaluate the benefits of yoga as a 'mind-body' practice, by measuring it's effects on health-related psychological and physiological variables. The study also aims to investigate whether an association exists between subjective (psychological) and objective (physiological) measures, with a particular focus on stress as the primary outcome.

DETAILED DESCRIPTION:
Stress and worry in everyday life are common features of Western society. Stress is a biological mechanism tapping the fight-or-flight-response via activation of the sympathetic nervous system. When exposed to stress during prolonged periods of time, the immune system is affected, leading to physiological as well as psychosocial problems. The consequences of untreated high stress can not only turn into reduced job capacity, and work roles conflicts, but also into cardiovascular disease, and mental illness such as an anxiety disorder or/and depression.

One common and recommended strategy to manage stress is to exercise regularly. Yoga is an umbrella term for a wide variety of physical, mental, and spiritual practices with its roots in ancient India. Most previous research on the health effects of yoga has demonstrated benefits on psychological health factors including mental stress, anxiety, depression and sleep problems.

The aim of the study is thus to investigate the effects of two types of yoga intervention on psychological and physiological health.

ELIGIBILITY:
Inclusion Criteria:

* A score on four items of the Perceived Stress Scale between 8-16, thereby indicating a current stress experience of at least moderate level.
* Ability to participate in the intervention during the time-period.
* Comprehensive in Swedish.

Exclusion Criteria:

* Ongoing yoga practice or any regular practice of yoga or meditation within the last 6 months.
* Any known physical limitations that may prevent light physical activity (yoga postures).
* Current psychological or psychopharmacological treatment.
* Inability to attend more than 5 of the scheduled 10 yoga sessions.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2016-04-23 (Actual); Study Completion 2016-04-23 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | 5 weeks
  A 10-item scale measuring the degree to which situations in one's life are appraised as stressful.The items are rated on a 5-point scale from 0 (never) to 4 (very often). Total scores range from 0 to 40, with higher scores indicating a higher stress level.
The Hospital Anxiety and Depression Scale | 5 weeks
  A fourteen item scale which assesses levels of anxiety and depression. Seven of the 14 items relate to anxiety and seven relate to depression. Each item is scored from 0-3. Items can be scored together by subscale (score range: 0-21), or for total scale score (score range: 0-42).
The COPE Inventory | 5 weeks
  Assesses 14 conceptually distinct coping strategies. It includes 13 scales with four items each and one single item question to assess different strategies for coping with stress. All items are reported on a 4-point scale.
The Insomnia Severity Index | 5 weeks
  A brief screening measure of insomnia and an outcome measure for use in intervention research. The index contains seven items rated on a five-point Likert scale from 0 to 4. Higher scores indicate symptoms of insomnia.
Diet | 5 weeks
  A 2-item measure that is used as an exploratory questionnaire. The questions are as follows: Have you changed your eating habits since you started your participation in the study? Categorical answer choices include 1) No, not at all, 2) Yes, to some extent, 3) Yes, to a great extent. A second question is open-ended: If you have changed your eating habits, please describe how. This very brief questionnaire will be given only once at the end of the study to explore whether dietary changes have occurred following the 5-week study period.
General Health Questionnaire | 5 weeks
  Consists of 12 items, each one assessing the severity of a mental problem over the past few weeks using a 4-point Likert-type scale (from 0 to 3). These scores generate a total score ranging from 0 to 36 where higher scores indicate worse health.
The Harmony in Life Scale | 5 weeks
  Assesses a global sense of harmony in one's life and consists of 5 statements for which participants are asked to indicate degree of agreement on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). The harmony score is established by summarizing the 5 statements for each participant, allowing for a maximum score of 35 (range: 5 - 35). Higher scores represent greater harmony in life.
The Kentucky Inventory of Mindfulness Skills -Short Version | 5 weeks
  A 20-item multi-dimensional scale of interrelated skills related to what one does while practicing mindfulness, and how one does it.
The Brief Experiential Avoidance Questionnaire | 5 weeks
  A questionnaire which consists of 15 items used to assess behavioral avoidance , distress aversion, procrastination, distraction/suppression, repression/denial, and distress endurance. Participants are asked to indicate degree of agreement on a 6-point Likert scale (1 = strongly disagree, 6 = strongly agree). The score is established by summing all items (score range: 15 - 90).
The Self-Compassion Scale | 5 weeks
  A 26-item measure with six subscales, tapping the construct of self-compassion. The subscales are self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. Scores of subscales are added together for a total score representative of the level of self-compassion.
Fasting blood sampling | 5 weeks
  A total of 3 tubes will be collected for each participant, amounting to a total of 65ml of blood per person. Blood analysis will include stress hormones, inflammatory biomarkers, metabolic profiling, cardiometabolic biomarkers, cholesterol, triglycerides, creatinine, catecholamines (noradrenalin and adrenalin), renin, cortisol, and glucose concentration.
Fasting and 120-minute glucose tolerance test (mmol/L) | 5 weeks
  The glucose tolerance test determines how the body responds to glucose (sugar). After a fasting blood sample is taken (see above procedure), participants will be asked to drink a liquid containing glucose. A second blood sample will be taken 120 minutes later.
Office and 24-hour blood pressure measurement (mmHg) | 5 weeks
  Blood pressure measurements will be taken periodically by the device for a period of 24-hours.
Pulse-wave velocity | 5 weeks
  Measured using a sphygmocor device.
Heart rate variability | 5 weeks
  Measured with electrocardiogram during deep breathing. Heart rate variability is is the variation in the time interval between heartbeats.
Gut microbiota | 5 weeks
  Fecal samples.

CONTACTS AND LOCATIONS:
Overall Officials: Olle Melander, MD, Prof., Principal Investigator — Lund University
Locations (1):
- KFE, Skåne University Hospital in Malmö, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daukantaite D, Tellhed U, Maddux RE, Svensson T, Melander O. Five-week yin yoga-based interventions decreased plasma adrenomedullin and increased psychological health in stressed adults: A randomized controlled trial. PLoS One. 2018 Jul 18;13(7):e0200518. doi: 10.1371/journal.pone.0200518. eCollection 2018. PMID 30020987

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT03428542/Prot_SAP_000.pdf